CLINICAL TRIAL: NCT00603122
Title: Acclimatization Mechanisms During Ascent to 7500m. Effects of Ascent Protocol on Acute Mountain Sickness and Cardiorespiratory Physiology
Brief Title: Acclimatization Mechanisms During Ascent to 7500m
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Konrad E. Bloch, University Hospital Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EK-1189; SNSF 3200B0-108300
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Acute Mountain Sickness
Keywords: altitude illness; hypoxia
MeSH Terms: conditions — Altitude Sickness; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): fast ascent
  Interventions: Behavioral: ascent protocol
- 2 (Active Comparator): slow ascent
  Interventions: Behavioral: ascent protocol

INTERVENTIONS:
Behavioral: ascent protocol — ascent protocol for the two groups has different acclimatization time

SUMMARY:
The trial evaluates the role of ascent protocol on acute mountain sickness and cardio-respiratory physiology during an ascent to Muztagh Ata (7546m). Two groups of mountaineers ascend with different acclimatization time to the summit. The prevalence and severity of symptoms of acute mountain sickness are evaluated along with physiologic variables.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, physically fit subject
* Mountaineering experience

Exclusion Criteria:

* Any type of cardiac or respiratory disease
* Regular intake of any medication
* History of high altitude pulmonary oedema
* Severe acute mountain sickness at altitudes below 3500m or high altitude cerebral oedema.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
acute mountain sickness | during ascent

SECONDARY OUTCOMES:
mountaineering success, oxygen saturation, breathing pattern | during ascent

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Principal Investigator — Pulmonary Division, University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Bloch KE, Latshang TD, Turk AJ, Hess T, Hefti U, Merz TM, Bosch MM, Barthelmes D, Hefti JP, Maggiorini M, Schoch OD. Nocturnal periodic breathing during acclimatization at very high altitude at Mount Muztagh Ata (7,546 m). Am J Respir Crit Care Med. 2010 Aug 15;182(4):562-8. doi: 10.1164/rccm.200911-1694OC. Epub 2010 May 4. PMID 20442435
- [Background] Garde A, Giraldo BF, Jane R, Latshang TD, Turk AJ, Hess T, Bosch MM, Barthelmes D, Hefti JP, Maggiorini M, Hefti U, Merz TM, Schoch OD, Bloch KE. Periodic breathing during ascent to extreme altitude quantified by spectral analysis of the respiratory volume signal. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:707-10. doi: 10.1109/EMBC.2012.6346029. PMID 23365990
- [Background] Latshang TD, Turk AJ, Hess T, Schoch OD, Bosch MM, Barthelmes D, Merz TM, Hefti U, Hefti JP, Maggiorini M, Bloch KE. Acclimatization improves submaximal exercise economy at 5533 m. Scand J Med Sci Sports. 2013 Aug;23(4):458-67. doi: 10.1111/j.1600-0838.2011.01403.x. Epub 2011 Nov 3. PMID 22093058
- [Result] Bloch KE, Turk AJ, Maggiorini M, Hess T, Merz T, Bosch MM, Barthelmes D, Hefti U, Pichler J, Senn O, Schoch OD. Effect of ascent protocol on acute mountain sickness and success at Muztagh Ata, 7546 m. High Alt Med Biol. 2009 Spring;10(1):25-32. doi: 10.1089/ham.2008.1043. PMID 19326598